CLINICAL TRIAL: NCT01587300
Title: N2004-05: Neuroblastoma Biology Study
Brief Title: Neuroblastoma Biology Study
Status: Recruiting | Type: Observational
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: N2004-05
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biospecimen includes blood and bone marrow and their derivatives (e.g., DNA, RNA, plasma, lymphocytes) as well as tumors.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Medical scientists want to find better ways to treat neuroblastoma and to find ways to prevent the tumor from growing back. To do this, they need more information about the characteristics of neuroblastoma cells. Therefore, they want to study samples of neuroblastoma tissues and neuroblastoma and normal cells in the blood and bone marrow that may be related to the growth of neuroblastoma cells. Doctors and other medical scientists also want to find better ways to detect and measure neuroblastoma to improve the ability to follow the response of tumor cells to therapy.

DETAILED DESCRIPTION:
The purposes of this study are:

To establish a storage place or bank of samples of blood, bone marrow, and/or tumor, and molecular components isolated from these samples from children with neuroblastoma. The stored specimens will be shared with laboratory researchers studying high risk neuroblastoma.

To collect clinical data (such as treatments received, date of diagnosis, tumor stage, etc) and radiology scans to provide this information as needed for the laboratory studies to be done on the specimens.

To obtain neuroblastoma tumor cells from tumor tissue, bone marrow, and/or blood to use to start cell lines, or tumor cells that will keep growing in the laboratory. These cell lines will be shared with laboratory researchers studying high risk neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be greater than or 31 days of age.
* Patients must have had a diagnosis of high risk neuroblastoma either by histological verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.
* All patients with refractory or recurrent high risk neuroblastoma at NANT institutions are eligible regardless of disease status (including no measurable or evaluable tumor) as long as they undergo a disease evaluation and appropriate samples are submitted.
* Additionally, all patients with high risk neuroblastoma without relapse treated at a NANT institution are eligible if undergoing a disease evaluation, as long as Children's Oncology Group specimens are prioritized.

Exclusion Criteria:

* There are no exclusion criteria on this study.

Ages: 31 Days to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neuroblastoma patients from various NANT sites.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-07; Primary Completion 2099-12 (Estimated); Study Completion 2099-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shahab Asgharzadeh, MD, Study Chair — Children's Hospital Los Angeles
Locations (17):
- United States (16):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucille Salter Packer Children's Hospital, Stanford University, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children Hospital of Colorado, Aurora, Colorado
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - University of Chicago, Comer Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - C.S Mott Children's Hospital, Ann Arbor, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada